CLINICAL TRIAL: NCT01397136
Title: Cell-free DNA: a Non-invasive Test for Assessing Embryo Quality
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Collaborators: Merck Serono S.A., Geneva (Industry)
Responsible Party: Principal Investigator, Paola Scaruffi, Dr, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Other Study IDs: GFI2011_PS
Record Dates: First submitted 2011-07-14; First posted 2011-07-19 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Culture Media; DNA
Keywords: Human embryo; Culture media; Cell-free DNA; In vitro fertilization; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After normally fertilized oocytes will be identified, they will be transferred into Sydney IVF Cleavage Medium (Cook Medical) for culture from day 1 to day 3 (up to 8 cell stage). For a subset of embryos we will also perform culture until blastocyst stage. For this purpose, embryos will be transferred into Sydney IVF Blastocist medium (Cook Medical) from day 3 to day 5/6. We will focus on embryo development in a single embryo culture medium. Embryos will be cultured at 37°C, 6.0% CO2, 5.0% O2 into Galaxy 48R incubators (New Brunswick Scientific). At the moment of transfer of embryos into the uterine cavity, we will collect embryo culture media into DNase- and RNase-free 1.5 ml tubes (Eppendorf AG). The media will be immediately frozen and stored at -20° until nucleic acid purification.
Oversight: Data Monitoring Committee: No

SUMMARY:
In the present project we propose to deeply characterize nuclear and/or mitochondrial DNA in embryo culture medium, in order to investigate whether both cell-free nucleic acid types may provide additional, reliable, predictive parameters for embryo viability and implantation potential.

ELIGIBILITY:
Inclusion Criteria:

* We will enroll in the study only embryos obtained from fresh gametes. It is to note that we currently transfer more than one embryo (with a maximum of 3, according to patient's age) and we will follow such criteria alongside the project. Consequently, we will take into consideration this aspect in correlating DNA parameters with embryo's outcome.

Exclusion Criteria:

* We will exclude cryopreserved embryos, in order to avoid potential biases due to cooling/defrosting procedures.

Ages: 2 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Culture media from human embryos collected at day 2-7 after in-vitro fertilization.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Isolation and characterization of nuclear and/or mitocondrial DNA into embryo culture medium | Month 6 of the project

SECONDARY OUTCOMES:
Prediction of high quality embryos according to molecular profiling of cell-free DNA released into culture medium. | Month 12 of the project
Publication of scientific reports. | Month 12 of the project
Dissemination of results by participating at national and international meetings, workshops and specific courses. | Months 3-12 of the project

CONTACTS AND LOCATIONS:
Overall Officials: Paola Scaruffi, PhD, Principal Investigator — UOS Physiopathology of Human Reproduction, IRCCS AOU San Martino-IST, Genoa, Italy
Locations (1):
- IRCCS AOU San Martino-IST, Genova, GE, Italy

REFERENCES:
- [Result] Stigliani S, Anserini P, Venturini PL, Scaruffi P. Mitochondrial DNA content in embryo culture medium is significantly associated with human embryo fragmentation. Hum Reprod. 2013 Oct;28(10):2652-60. doi: 10.1093/humrep/det314. Epub 2013 Jul 25. PMID 23887072
- [Result] Stigliani S, Persico L, Lagazio C, Anserini P, Venturini PL, Scaruffi P. Mitochondrial DNA in Day 3 embryo culture medium is a novel, non-invasive biomarker of blastocyst potential and implantation outcome. Mol Hum Reprod. 2014 Dec;20(12):1238-46. doi: 10.1093/molehr/gau086. Epub 2014 Sep 17. PMID 25232043